CLINICAL TRIAL: NCT04658160
Title: Longitudinal Tracking and Intervention Platform for Medicare Advantage Patients: A Prospective RCT
Brief Title: Longitudinal Tracking and Intervention Platform for Medicare Advantage Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Robin Kamal, Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 59260
Record Dates: First submitted 2020-12-01; First posted 2020-12-08 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Frailty
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): None- normal care
- Intervention/Tracking (Experimental): This group will have access to the longitudinal tracking and intervention platform for Medicare Advantage patients. Members of this group's care team will have access to the longitudinal data on the platform and will be able to intervene if any red flags emerge (i.e. if a patient displays signs of depression on a patient reported outcome measure/survey)
  Interventions: Behavioral: Longitudinal Tracking and Intervention Platform for Medicare Advantage Patients

INTERVENTIONS:
Behavioral: Longitudinal Tracking and Intervention Platform for Medicare Advantage Patients — access to/use of the tracking platform
  Arms: Intervention/Tracking

SUMMARY:
This study investigates whether a health tracking platform improves an elderly person's health with regards to frailty over the course of a year. Secondary research questions examine which instruments are the best predictors of frailty to improve preventative measures in the future.

DETAILED DESCRIPTION:
All patients presenting to the Annual Wellness Visit at Stanford Hospital will be considered for this study. Eligible who consent will be asked to conduct several activities, which will be video taped and timed.

The activities include:

* Timed up and go: patients will be asked to rise from a chair and walk 10 feet (3 m), turn, walk back to the chair, and sit down.
* QuickDASH tasks: open a jar, carry a shopping bag, cut food with a knife, wash back, wash a wall, and hammer a piece of wood.
* KOOS JR tasks: go up/down stairs, stand upright
* PROMIS PF tasks: lift heavy object repeat x5, shoelace or buttons, wash hair

Patients will then be asked to complete a survey consisting of a number of validated questionnaires used to collect patient reported outcome measures and assess frailty. Patients will be randomly assigned to one of two conditions, the control condition or the frailty wellness platform condition. Patients assigned to the frailty wellness platform condition will be given an orientation to a health tracking program. They will be asked to fill out the questionnaires at 3 separate time points on the program site (accessed via phone or computer) at 3 months, 6 months, and 9 months, following orientation. One year later, at the patient's second Annual Wellness Visit, the patient will be asked to fill out the Health Risk Assessment and the study will conclude.

ELIGIBILITY:
Inclusion Criteria:

* geriatric patients >65 years of age

Exclusion Criteria:

* none

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Health Risk Assessment | Change in participant's Health Risk Assessment from beginning of study to end (1 year duration)
  A multi-component health survey representing the participant's assessment of their health status

CONTACTS AND LOCATIONS:
Overall Officials: Robin Kamal, MD MBA, Principal Investigator — Stanford University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morley JE, Malmstrom TK, Miller DK. A simple frailty questionnaire (FRAIL) predicts outcomes in middle aged African Americans. J Nutr Health Aging. 2012 Jul;16(7):601-8. doi: 10.1007/s12603-012-0084-2. PMID 22836700
- [Background] Liu LH, Garrett SB, Li J, Ragouzeos D, Berrean B, Dohan D, Katz PP, Barton JL, Yazdany J, Schmajuk G. Patient and clinician perspectives on a patient-facing dashboard that visualizes patient reported outcomes in rheumatoid arthritis. Health Expect. 2020 Aug;23(4):846-859. doi: 10.1111/hex.13057. Epub 2020 Apr 9. PMID 32270591